CLINICAL TRIAL: NCT04302766
Title: Intermediate-Size Patient Population Expanded Access Treatment Protocol for Coronavirus Disease 2019 (COVID-19) Remdesivir (RDV; GS-5734™)
Brief Title: Expanded Access Remdesivir (RDV; GS-5734™)
Status: No longer available | Type: Expanded Access
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: S-20-01
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19; GS-5734; Remdesivir; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Remdesivir — Remdesivir (RDV,GS-5734) is a monophosphoramidate prodrug of an adenosine analog with potent activity against an array of RNA virus families including Filoviridae, Paramyxoviridae, Pneumoviridae, and Orthocoronavirinae, through the targeting of the viral RNA dependent RNA polymerase (RdRp).
  Other Names: GS-5734

SUMMARY:
Disease caused by 2019 Novel Coronavirus also known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)

DETAILED DESCRIPTION:
The treatment of communicable Novel Coronavirus (CODIV-19) of 2019 with Remdesivir (RDV; GS-5734™) also known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)

ELIGIBILITY:
Inclusion Criteria:

* DoD-affiliated personnel as defined in DoDI 6200.02, which includes emergency-essential civilian employees and/or contractor personnel accompanying the Armed Forces who are subject to the same health risk as military personnel
* Have a laboratory-confirmed COVID-19 diagnosis with moderate to severe disease presentation as determined by the principal investigator
* Patient or legally authorized representative (LAR) provides written informed consent, except as noted in 21 CFR 50.23
* Understands and agrees to comply with planned study procedures
* Available for clinical follow-up for duration of the treatment and follow-up period
* Woman of childbearing potential must

  * Have a negative pregnancy test within 24 hours before starting treatment
  * Agree not to become pregnant during treatment and for 1 months after receiving remdesivir (Treatment will be a maximum of 10 doses given over a 10-day interval)
  * Use at least 2 reliable forms of effective contraception, including 1 barrier method, during treatment and for 1 month after the treatment period

Exclusion Criteria:

* ALT/AST ≥ 5 times the upper limit of normal
* Stage 4 severe kidney disease or requiring dialysis (i.e. eGFR <30)
* Anticipated transfer to another hospital that is not a study site within 72 hours
* Allergy to any components of the study medication [GS-5734, sulfobutylether β-cyclodextrin sodium (SBECD) and hydrochloric acid and/or sodium hydroxide]
* Concomitant antiviral therapy (lopinavir/ritonavir [Kaletra])
* Pregnant or nursing

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (14):
  - Naval Medical Center San Diego, San Diego, California
  - Naval Hospital Jacksonville, Jacksonville, Florida
  - Benning Martin Army Community Hospital, Fort Benning, Georgia
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Tripler Army Medical Center, Tripler AMC, Hawaii
  - Blanchfield Army Community Hospital, Fort Campbell North, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Naval Medical Center Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina
  - William Beaumont Army Medical Center, El Paso, Texas
  - Carl R. Darnall Army Medical Center, Fort Hood, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
- Afghanistan (2):
  - Craig Joint Theater Hospital, Bagrām
  - NATO Role 3 Multinational Medical Unit Kandahar Air Field, Kandahar
- EMF Camp Lemonnier, Djibouti, Djibouti
- Landstuhl Regional Medical Center, Landstuhl, APO AE, Germany
- US Naval Hospital Guam, Hagåtña, Guam
- Baghdad Diplomatic Support Center, Baghdad, Iraq
- US Naval Hospital Okinawa, Okinawa, Japan
- US Military Hospital Kuwait 411th Hospital Center, Kuwait City, Kuwait

DOCUMENTS (1):
  • Informed Consent Form (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT04302766/ICF_000.pdf